CLINICAL TRIAL: NCT01593280
Title: Quality of Recovery Following Administration of Transverse Abdominus Plane (TAP) Catheter as Compared to Intrathecal Morphine After Cesarean Delivery Under Spinal Anesthesia: a Prospective, Randomized Trial
Brief Title: TAP Catheters Versus Intrathecal Morphine for Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stamford Anesthesiology Services, PC (Other)
Collaborators: I-Flow (Industry)
Responsible Party: Principal Investigator, Dr. Vlad Frenk, attending anesthesiologist, Stamford Anesthesiology Services, PC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0308.01
Record Dates: First submitted 2012-04-30; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Abdominal Muscles/Ultrasonography; Adult; Anesthetics, Local/Administration & Dosage; Ropivacaine/Administration & Dosage; Ropivacaine/Analogs & Derivatives; Cesarean Section; Humans; Nerve Block/Methods; Pain Measurement/Methods; Pain, Postoperative/Prevention & Control; Ultrasonography, Interventional
Keywords: anesthesia; regional anesthetic techniques: transversus abdominis plane block,; pain, postoperative; surgery, cesarean section; quality of recovery
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP catheter (Active Comparator): Indwelling TAP catheter placed at the end of c-section. It will be dosed with 20ml of Ropivacaine 0.5% at that time. Double lumen OnQ C-block pump containing 700 ml of the Ropivacaine 0.2% will be attached to the TAP catheters in the recovery room. The catheters will run at 7cc/hr/side for 50 hrs.
  Interventions: Device: TAP catheter
- intrathecal morphine (Active Comparator): 0.3 mg of intrathecal morphine
  Interventions: Drug: intrathecal morphine

INTERVENTIONS:
Device: TAP catheter — dosed with 20ml of Ropivacaine 0.5% at that time. Double lumen pump containing 700 ml of the Ropivacaine 0.2% will be attached to the TAP catheters in the recovery room. The time that this occurs will be recorded in the eMAR. The catheters will run at 7cc/hr/side for 50 hrs.
  Other Names: On Q pump
  Arms: TAP catheter
Drug: intrathecal morphine — 0.3 mg
  Other Names: Duramorph
  Arms: intrathecal morphine

SUMMARY:
Morphine, when given as part of spinal anesthesia, is associated high incidence of nausea and pruritus, which may affect quality of recovery. The investigators hypothesize that long-acting local anesthetic infusions via TAP catheter can provide better quality of recovery after cesarean section than spinal morphine.

DETAILED DESCRIPTION:
This study is a prospective, open, randomized study. Subjects will be randomized using a computer-generated table of random numbers into 2 groups. The first group will receive intrathecal morphine as part of a spinal anesthetic. The second group will receive an ultrasound-guided bilateral TAP catheter at the end of the procedure, while the subject is still under the effect of spinal anesthetic. Group assignments will be sealed in sequentially numbered, opaque envelopes that would be opened by an anesthesiologist performing the cesarean section. The research nurse or one of the investigators, not involved with patient care after the subject signed written informed consent, will provide postoperative data collection.

All patients will be pre-hydrated with 1000ml of Lactated Ringer's solution. They will then be brought to the OR and without premedication receive a spinal anesthetic in a sitting position. The spinal anesthetic will be administered at either L3-4 or L4-5 level with 24G Sprotte needle and contain 1.4ml of 0.75% hyperbaric bupivacaine. As per protocol, the first group would receive 0.3mg of preservative-free morphine, mixed in the same syringe. All the subjects then will be immediately placed in supine position with left uterine displacement, and supplemental oxygen 4L/min will be administered via nasal cannula for the duration of procedure. After a successful spinal anesthetic is confirmed by loss of sensation to pinprick, cesarean section will be performed. Intraoperative hypotension will be treated with IV fluids, as well as intermittent boluses of IV ephedrine or IV neosynephrine as needed to keep SBP>100mm Hg. Intraoperative nausea will be treated with IV ondansetron as needed.

At the end of the procedure, the second group will receive ultrasound guided TAP catheter using a linear 6-15MHz ultrasound probe on a portable ultrasound machine (SonoSite, Bothell, WA) as previously described (Hebbard P, 2007). Each catheter will be dosed with 20ml of Ropivacaine 0.5% at that time. Double lumen OnQ C-block pump (I-Flow, LLC, Lake Forest, CA) containing 700 ml of the Ropivacaine 0.2% will be attached to the TAP catheters in the recovery room. The time that this occurs will be recorded in the eMAR. The catheters will run at 7cc/hr/side for 50 hrs.

In the recovery area, the patient will be asked to rate their pain at rest, nausea, and pruritus upon arrival and at regular intervals as per routine care. The pain will be rated on a 0 to 10 numeric rating scale (NRS), where 0 means no pain and 10 is the worst pain imaginable. Fentanyl 50 mg IV will be administered every 5 minutes to maintain an NRS pain score <4 of 10. Nausea will be rated on a 0 to 2 scale (0 = no nausea and vomiting, 1 = mild to moderate nausea or vomiting not needing treatment, and 2 = severe nausea or vomiting needing treatment). It will be treated with 4mg IV ondansetron, if necessary. The presence of pruritus and whether the treatment is desired will be assessed on a 0 to 2 scale (0= no pruritus, 1= mild pruritus not requiring treatment, 2= moderate pruritus requiring treatment or severe pruritus). Pruritus will be treated with IV diphenhydramine 25 mg if the subject weighs less than 150lbs and 50mg if the subjects weighs more than 150lbs. Upon transfer to the maternity floor, the nurses will ask the subjects to rate their pain at rest, nausea, and pruritus as part of usual care, upon arrival and every 4 hours for 48 hours as described above. The answers will be recorded on a data collection too. For the following 48 hours, the patient will be treated as follows: nausea will be treated with 25 mg IV promethazine followed by 4mg IV ondansetron if necessary every 6 hours. Pruritus will be treated with IV/PO diphenhydramine 25 mg if the subject weighs less than 150lbs and 50mg if the subject weighs more than 150lbs every 6 hours if necessary. Pain will be treated with SQ morphine (4mg for NRS pain 3-4, 6 mg for NRS pain 4-7, 8mg for NRS pain >7) every 4 hours as requested and 30mg IV ketorolac every 6 hours until subjects start eating. Once the subject tolerate diet, their pain will be treated with 800 mg PO ibuprofen every 6 hours and a combination of oxycodone 5mg and acetaminophen 325mg PO every 4 hours as requested (1 tab for NRS pain 4-7, 2 tabs for NRS pain >7).

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 - 45 years of age undergoing cesarean section under spinal anesthesia.
* Ability to read and write English

Exclusion Criteria:

* Patients undergoing other concomitant procedure
* Patients with history of diabetes or chronic steroid use
* Patients with chronic or recent (within 1 week prior to procedure) opioid use.
* Patients without the mental capacity to consent for the procedure/study.
* Patients requiring a translator in order to sign the consent for the procedure/study.
* Patients with a history of allergic reactions to local anesthetics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery after cesarean section | 48 hours
  To determine whether using continuous TAP catheters would result in a better quality of recovery after elective cesarean section under spinal anesthesia as compared to intrathecal morphine using QoR-40 questionnaire

SECONDARY OUTCOMES:
Incidence of nausea/vomiting | 48 hours
  nausea scores (0-2) and daily dose of antiemetic
incidence and severity of pruritus | 48 hours
  pruritis on 0-2 scale. Daily dose of antipruritic medications
overall oral narcotic use during the 48 hours post-operatively | 48 hours
  Postoperative data collection will include pain scores (0-10) and daily oral narcotic use

CONTACTS AND LOCATIONS:
Locations (1):
- Stamford Hospital, Stamford, Connecticut, United States

REFERENCES:
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Loane H, Preston R, Douglas MJ, Massey S, Papsdorf M, Tyler J. A randomized controlled trial comparing intrathecal morphine with transversus abdominis plane block for post-cesarean delivery analgesia. Int J Obstet Anesth. 2012 Apr;21(2):112-8. doi: 10.1016/j.ijoa.2012.02.005. Epub 2012 Mar 10. PMID 22410586
- [Background] Eslamian L, Jalili Z, Jamal A, Marsoosi V, Movafegh A. Transversus abdominis plane block reduces postoperative pain intensity and analgesic consumption in elective cesarean delivery under general anesthesia. J Anesth. 2012 Jun;26(3):334-8. doi: 10.1007/s00540-012-1336-3. Epub 2012 Feb 22. PMID 22354671
- [Background] McMorrow RC, Ni Mhuircheartaigh RJ, Ahmed KA, Aslani A, Ng SC, Conrick-Martin I, Dowling JJ, Gaffney A, Loughrey JP, McCaul CL. Comparison of transversus abdominis plane block vs spinal morphine for pain relief after Caesarean section. Br J Anaesth. 2011 May;106(5):706-12. doi: 10.1093/bja/aer061. PMID 21498494
- [Background] Costello JF, Moore AR, Wieczorek PM, Macarthur AJ, Balki M, Carvalho JC. The transversus abdominis plane block, when used as part of a multimodal regimen inclusive of intrathecal morphine, does not improve analgesia after cesarean delivery. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):586-9. doi: 10.1097/aap.0b013e3181b4c922. PMID 19916252
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] Charuluxananan S, Kyokong O, Somboonviboon W, Narasethakamol A, Promlok P. Nalbuphine versus ondansetron for prevention of intrathecal morphine-induced pruritus after cesarean delivery. Anesth Analg. 2003 Jun;96(6):1789-1793. doi: 10.1213/01.ANE.0000066015.21364.7D. PMID 12761013
- [Background] De Oliveira GS Jr, Fitzgerald PC, Marcus RJ, Ahmad S, McCarthy RJ. A dose-ranging study of the effect of transversus abdominis block on postoperative quality of recovery and analgesia after outpatient laparoscopy. Anesth Analg. 2011 Nov;113(5):1218-25. doi: 10.1213/ANE.0b013e3182303a1a. Epub 2011 Sep 16. PMID 21926373
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Liu SS, Wu CL. The effect of analgesic technique on postoperative patient-reported outcomes including analgesia: a systematic review. Anesth Analg. 2007 Sep;105(3):789-808. doi: 10.1213/01.ane.0000278089.16848.1e. PMID 17717242